CLINICAL TRIAL: NCT02871739
Title: A Pilot Randomized Trial Comparing Approaches to Shared Decision Making Skills Training for Clinicians
Brief Title: A Trial Comparing Approaches to Shared Decision Making Skills Training for Clinicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Partners HealthCare (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Director Health Decision Sciences Center, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016P000470
Record Dates: First submitted 2016-08-09; First posted 2016-08-18 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: Depression; Low Back Pain
Keywords: Communication skills training; Shared Decision Making; Decision making; Decision Aids; lung cancer screening
MeSH Terms: conditions — Depression; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- DA viewing with SPI Feedback (Experimental): Group 1 receives three decision aids and feedback on their standardized patient (SPI) interaction rating their shared decision making skills and highlighting opportunities for improvement.
  Interventions: Behavioral: DA viewing; Behavioral: SPI feedback
- DA viewing with no SPI Feedback (Experimental): Group 2 receives three decision aids. This group does not receive any feedback from the SPI.
  Interventions: Behavioral: DA viewing
- Webinar with SPI Feedback (Experimental): Group 3 receives an online, interactive webinar that focuses on SDM skills in clinical encounters and feedback on their standardized patient (SPI) interaction rating their shared decision making skills and highlighting opportunities for improvement.
  Interventions: Behavioral: Webinar; Behavioral: SPI feedback
- Webinar with no SPI Feedback (Experimental): Group 4 receives an online, interactive webinar that focuses on SDM skills in clinical encounters. This group does not receive any feedback from the SPI.
  Interventions: Behavioral: Webinar

INTERVENTIONS:
Behavioral: Webinar — 1 hour online, interactive webinar that covers shared decision making skills in clinical encounters.
  Arms: Webinar with SPI Feedback; Webinar with no SPI Feedback
Behavioral: DA viewing — Participants will receive 3 decisions aids to review.
  Arms: DA viewing with SPI Feedback; DA viewing with no SPI Feedback
Behavioral: SPI feedback — Rating of shared decision making skills and opportunities for improvement based on transcript of a standardized patient interaction
  Arms: DA viewing with SPI Feedback; Webinar with SPI Feedback

SUMMARY:
The Health Decision Sciences Center (HDSC) staff has deployed different approaches to training clinicians to engage patients in shared decision making for common medical tests and treatments. The purpose of the study is to compare the effectiveness of shared decision making (SDM) skills training courses using standardized patient interactions (SPI) and written evaluations.

DETAILED DESCRIPTION:
There is limited evidence on approaches to training clinicians to engage patients in shared decision making for common medical tests and treatments. The purpose of the study is to compare the effectiveness of different approaches to shared decision making (SDM) skills training. Participants will be randomly assigned to either receive two decision aids or a webinar to review. Participants will also be randomly assigned to receive feedback on standardized patient interaction rating their shared decision making skills and highlighting opportunities for improvement or not. Clinician participants will be assigned to one of four intervention groups using a 2x2 factorial design:

Group 1: Decision aid viewing with feedback Group 2: Decision aid viewing and no feedback Group 3: webinar with feedback Group 4: webinar and no feedback

The pilot study will provide evidence on the comparative effectiveness and feasibility on training formats to determine if:

* Clinicians improved in SDM communication skills
* Clinicians have an increased confidence to use SDM with their patients
* The training is acceptable to clinicians

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 and older
* English speaking
* Physician
* Nurse Practitioner
* Physician Assistant
* Registered Nurse

Exclusion Criteria:

* Not clinically active (research faculty only)
* Medical Trainees
* Medical Students
* Medical Assistants
* Social Workers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sepucha, PhD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Legare F, Stacey D, Turcotte S, Cossi MJ, Kryworuchko J, Graham ID, Lyddiatt A, Politi MC, Thomson R, Elwyn G, Donner-Banzhoff N. Interventions for improving the adoption of shared decision making by healthcare professionals. Cochrane Database Syst Rev. 2014 Sep 15;(9):CD006732. doi: 10.1002/14651858.CD006732.pub3. PMID 25222632
- [Background] Davis D. Does CME work? An analysis of the effect of educational activities on physician performance or health care outcomes. Int J Psychiatry Med. 1998;28(1):21-39. doi: 10.2190/UA3R-JX9W-MHR5-RC81. PMID 9617647
- [Background] Price EL, Bereknyei S, Kuby A, Levinson W, Braddock CH 3rd. New elements for informed decision making: a qualitative study of older adults' views. Patient Educ Couns. 2012 Mar;86(3):335-41. doi: 10.1016/j.pec.2011.06.006. Epub 2011 Jul 14. PMID 21757315

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DA Viewing With SPI Feedback | DA Viewing With no SPI Feedback | Webinar With SPI Feedback | Webinar With no SPI Feedback
Started | 6 | 6 | 4 | 7
Completed First SPI | 3 | 5 | 4 | 6
Completed Second SPI | 3 | 4 | 4 | 5
Complete Final Survey | 3 | 4 | 4 | 5
Completed | 3 | 4 | 4 | 5
Not Completed | 3 | 2 | 0 | 2
Not completed — Lost to Follow-up | 3 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DA Viewing With SPI Feedback | DA Viewing With no SPI Feedback | Webinar With SPI Feedback | Webinar With no SPI Feedback | Total
Number analyzed (Participants) | 6 | 6 | 4 | 7 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 4 | 7 | 22
  >=65 years | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 4 | 6 | 17
  Male | 1 | 4 | 0 | 1 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 4 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Braddock's Informed Decision Making Score
Description: Transcripts from standardized patient interactions (SPI) will be scored using Braddock's Informed Decision Making (IDM) framework to assess shared decision making skills. Scores with the Braddock's Informed Decision Making Framework range from 0 to 9; the higher scores are better. We subtracted the scores of the baseline SPI collected before the intervention from the second SPI collected 4-6 weeks later, after the intervention, to determine the change in IDM score for each participant and then compared change scores across study arms.
Time Frame: Baseline (before intervention) and 4-6 weeks (after intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DA Viewing With SPI Feedback | DA Viewing With no SPI Feedback | Webinar With SPI Feedback | Webinar With no SPI Feedback
Number analyzed (Participants) | 3 | 4 | 4 | 5
score on a scale | 2.00 (1.29) | 1.25 (2.06) | 1.00 (0.82) | 3.20 (1.79)

ADVERSE EVENTS:
Time Frame: Serious and other (not including serious) adverse events were not collected/assessed.
Description: Adverse events were not collected.
Arm/Group | DA Viewing With SPI Feedback | DA Viewing With no SPI Feedback | Webinar With SPI Feedback | Webinar With no SPI Feedback
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes